CLINICAL TRIAL: NCT01052194
Title: A 12-week, Double-blind, Randomized, Parallel-group, Placebo-controlled Study of 4 Doses of VX-509 in Subjects With Active Rheumatoid Arthritis
Brief Title: A 12-week Study of 4 Doses of VX-509 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX09-509-101; 2009-017438-32 (EudraCT Number)
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 25 mg b.i.d. VX-509 (Experimental)
  Interventions: Drug: VX-509
- 50 mg b.i.d. VX-509 (Experimental)
  Interventions: Drug: VX-509
- 100 mg b.i.d. VX-509 (Experimental)
  Interventions: Drug: VX-509
- 150 mg b.i.d. VX-509 (Experimental)
  Interventions: Drug: VX-509
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — tablet, placebo b.i.d. for 12 weeks
  Arms: Placebo
Drug: VX-509 — tablets, 25mg b.i.d. for 12 weeks
  Arms: 25 mg b.i.d. VX-509
Drug: VX-509 — tablet, 50 mg b.i.d. for 12 weeks
  Arms: 50 mg b.i.d. VX-509
Drug: VX-509 — tablet, 100 mg b.i.d. for 12 weeks
  Arms: 100 mg b.i.d. VX-509
Drug: VX-509 — tablet, 150 mg b.i.d. for 12 weeks
  Arms: 150 mg b.i.d. VX-509

SUMMARY:
This study is designed to evaluate safety and assess initial efficacy of VX-509, a JAK3 inhibitor, for treatment of subjects with active RA. This study will assess the clinical response of 4 doses of VX-509 compared to placebo when administered for 12 weeks to patients with active RA. The study will also evaluate the safety and tolerability of VX-509 compared to placebo when administered for 12 weeks to subjects with active RA.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have been diagnosed with RA as defined by the ACR revised criteria with disease duration of at least 6 months from confirmed diagnosis
* Subjects must have a swollen joint count of ≥6 out of 28 joints and tender joint count of ≥6 out of 28 joints. Joints that have had prior surgery are to be excluded from the joint count.
* Baseline CRP level must be 1.5 times greater than the upper limit of normal at Screening.
* Subjects must have failed at least 1 nonbiologic DMARD for any reason.
* Subjects may have previously failed no more than 1 biologic DMARD and discontinued treatment for reasons other than inadequate response. Subjects must not have been treated with Rituximab previously.
* Subjects must be willing to comply with contraception requirements.

Exclusion Criteria:

* Subjects with inflammatory rheumatological disorders other than RA.
* History or evidence of a clinically significant disorder other than RA (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric disorders), condition or disease that, in the opinion of the investigator and medical monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subjects with clinically important abnormalities in screening physical examination or in screening laboratory test results (including the presence of either hepatitis B surface antigen, hepatitis C virus antibody, or HIV types 1 -- Subjects with elevation in alanine aminotransferase or aspartate aminotransferase above the upper limit of normal.
* History of hematologic disorders including neutropenia and thrombocytopenia.
* Subjects with an acute or chronic active infection requiring systemic antimicrobial treatment, or subjects who are at high risk of developing an infection due to a compromised immune system. Antifungals for onychomycosis or low-dose antibiotics for rosacea, that are not inhibitors or inducers of CYP3A, will be allowed.
* Subjects who require concomitant use of any inhibitors or inducers of cytochrome P450 (CYP) 3A.
* Subjects who have been treated with intra-articular injections of corticosteroids within 28 days prior to Day 1.
* Subjects who have planned major surgery (e.g., joint replacement) or any procedures during the study.
* Have received any live, attenuated vaccinations within 1 month prior to study drug administration.
* History of drug or alcohol abuse or excessive alcohol as determined by the investigator, during the last 12 months before the screening visit.
* History of TB infection of any kind (pulmonary or extrapulmonary, active or latent), regardless of history of anti-TB treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve an ACR20 response | Week 12
Change from baseline in DAS28 | Week 12

SECONDARY OUTCOMES:
Proportion of subjects who achieve an ACR50,70 response | Week 12
Proportion of subjects who achieve moderate or good EULAR response | Week 12
Magnitude of improvement in the components of the ACR response criteria | Week 12
Pharmacokinetics of VX-509 | Week 6
Pharmacodynamics (PD) of biomarker responses | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (47):
- United States (17):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Peoria, Arizona
  - La Mesa, California
  - Trumbull, Connecticut
  - Tampa, Florida
  - Venice, Florida
  - Decatur, Georgia
  - Worcester, Massachusetts
  - St Louis, Missouri
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Spokane, Washington
  - Clarksburg, West Virginia
- Antwerp, Belgium
- Croatia (3):
  - Karlovac
  - Opatija
  - Zagreb
- Germany (6):
  - Erfurt
  - Frankfurt
  - Hamburg
  - Hildesheim
  - Nauheim
  - Zerbst
- Hungary (4):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Veszprém
- Poland (4):
  - Elblag
  - Limanow
  - Lublin
  - Wroclaw
- San Juan, Puerto Rico
- Romania (4):
  - Baia Mare
  - Brăila
  - Bucharest
  - Galati
- Russia (5):
  - Kemerovo
  - Novosibirsk
  - Ryazan
  - Vladimir
  - Voronezh
- Serbia (2):
  - Belgrade
  - Niška Banja